CLINICAL TRIAL: NCT06140537
Title: Efficacy and Mechanisms of Dapagliflozin in Promoting Kidney Function and Cardiovascular Health in Kidney Transplant Recipients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-1360
Record Dates: First submitted 2023-11-14; First posted 2023-11-20 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Kidney Transplant; Complications; Vascular Diseases; Diabetes
MeSH Terms: conditions — Vascular Diseases; Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dapagliflozin (Experimental): Participants will receive dapagliflozin 10mg daily
  Interventions: Drug: Dapagliflozin 10mg Tab
- Placebo (Placebo Comparator): Participants will receive one placebo tablet daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapagliflozin 10mg orally daily
  Arms: Dapagliflozin
Drug: Placebo — Placebo one tablet orally daily
  Arms: Placebo

SUMMARY:
Long-term allograft function in kidney transplant recipients (KTRs) remain suboptimal, and graft failure causes significant morbidity and mortality, with cardiovascular disease being the leading cause of death in KTRs and the most common cause of death with a functioning graft. Sodium-glucose cotransporter 2 (SGLT2) inhibitors safely lower cardiovascular and kidney disease risk in the non-transplant population, yet data in KTRs are lacking. This clinical trial seeks to establish the efficacy and safety of dapagliflozin, a SGLT2 inhibitor, for improving cardiovascular and kidney graft function in adult KTRs with type 2 diabetes and post-transplant diabetes, and to leverage innovate translational methods to define the underlying mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Kidney transplant received 1 year prior to randomization
* estimated glomerular filtration rate 30-90 ml/min/1.73m2
* Urine albumin to creatinine ratio (ACR) 30-5000 mg/g
* Pre-existing type 2 diabetes or post-transplant diabetes mellitus
* Blood pressure <130/80 mm Hg prior to randomization
* Able to provide informed consent
* Stable immunosuppression for at least 3 months prior to baseline consisting of tacrolimus, mycophenolate mofetil/mycophenolic acid and prednisone
* Stable anti-hypertensive regimen for at least 1month prior to baseline
* Stable diabetes management for at least 3 months prior to baseline
* Stable angiotensin converting enzyme inhibitor/angiotensin receptor blocker use for at least 3 months prior to baseline (if applicable)
* Glucagon-like peptide-1 receptor agonist (GLP-1RA) for at least 3 months prior to baseline (if applicable)

Exclusion Criteria:

* Type 1 diabetes
* Anticipated life expectancy <1 year
* Uncontrolled hypertension
* Hemoglobin A1c >9%
* Body mass index >40 kg/m2
* New York Heart Association Class 3 or 4 heart failure symptoms, an EF ≤30%, or hospitalization for heart failure in the past 3 months
* Pregnancy, plans to become pregnant, or breastfeeding
* Current use of sodium glucose cotransporter-2 (SGLT2) inhibitors
* Current urinary or urogenital infection
* Use of anticoagulants (contraindication to kidney biopsy)
* Magnetic resonance imaging (MRI) contraindications
* History of lower-limb amputation irrespective of etiology
* Known hypersensitivity to dapagliflozin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Albuminuria | Change from baseline to 12 months
  Measured by urine albumin to creatinine ratio

SECONDARY OUTCOMES:
Kidney fibrosis | Change from baseline to 12 months
  Measured by Magnetic Resonance Imaging (MRI) and kidney biopsy tissue
Kidney oxygenation | Change from baseline to 12 months
  Measured by MRI
Arterial stiffness | Change from baseline to 12 months
  Measured by aortic pulse wave velocity
Left ventricular mass | Change from baseline to 12 months
  measured by cardiac MRI
estimated glomerular filtration rate | Change from baseline to 12 months
  estimated by CKD epi equation
Kidney morphometry, metabolomics from paired kidney biopsies | Change from baseline to 12 months
  measured by single cell RNA sequencing from paired kidney biopsies
safety and tolerability | baseline, 6 and 12 months
  assessed on basis of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the study, data, which has been stripped of all personal identification information and coded with a number, will be made available to qualified individuals within the scientific community who apply for data use. The results and outcomes of this study will be made generally available by publication and journal articles submitted to PubMed Central in compliance with NIH access guidelines.
Supporting Information: Study Protocol, SAP
Time Frame: At the conclusion of the study, data, which has been stripped of all personal identification information and coded with a number, will be made available to qualified individuals within the scientific community who apply for data use. The results and outcomes of this study will be made generally available by publication and journal articles submitted to PubMed Central in compliance with NIH access guidelines.